CLINICAL TRIAL: NCT05678868
Title: Implementation of a Structural Mitral Valve Clinic for the Management of Patients With Heart Failure Refractory to Medical Therapy
Brief Title: Structural Mitral Valve Project
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Queen's University (Other)
Collaborators: AFP Innovation Fund (Other)
Responsible Party: Principal Investigator, Wael Abuzeid, MD, MSc, Interventional Cardiologist, Assistant Professor, Department of Medicine, Queen's University
Other Study IDs: Version Date January 25, 2022
Record Dates: First submitted 2022-09-07; First posted 2023-01-10 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2022-12

CONDITIONS: Mitral Regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: MitraClip procedure — MitraClip is surgical procedure to repair the mitral valve in your heart. During the procedure, the doctor will access the mitral valve using a thin tube (called a catheter) that is guided through a vein in your leg to reach your heart. A small implanted clip is attached to the mitral valve to reduce the leaking across the valve and to reduce symptoms and stress on the heart.

SUMMARY:
This is a prospective Quality Improvement (QI) study using the Model for Improvement framework.

The objective of this study is to implement a structured, comprehensive, innovative, and sustainable approach to the management of patients with advanced mitral valve (MV) disease and heart failure (HF) in Southeastern Ontario and to improve healthcare delivery, patient care, and patient outcomes in the context of structural surgical and percutaneous MV interventions. This will be achieved through the strategic implementation, promotion, and evaluation of:

i.The first local Southeastern Ontario Structural Mitral Valve Clinic using an Interdisciplinary heart team (IHT) at the Kingston Health Sciences Centre (KHSC) and its integration with the KHSC's existing Heart Failure Clinic; ii.The first provincial Structural Mitral Valve Clinic electronic referral service on the Ontario electronic services platform; and iii.The promotion of the above through targeted KT (Knowledge Transfer) outreach activities.

Patients for this study will be recruited through medical referral within the south eastern Ontario, Canada region.

ELIGIBILITY:
Inclusion Criteria:

All adults (≥18 years of age) patients with primary and secondary moderate to severe MR with HF (preserved or reduced ejection fraction with New York Heart Association (NYHA) Class >II), who have had at least one previous hospitalization for HR, require specialist advisement, and have provided signed informed consent.

Exclusion Criteria:

* Those who are not eligible for either an MV surgical intervention or a TMVI procedure.
* Females of childbearing age who are not willing or unable to use a reliable method of birth control.
* Inpatient referrals.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with primary and secondary moderate to severe MR with heart failure (HF) (preserved or reduced ejection fraction with New York Heart Association (NYHA) Class >II), who have had at least one previous hospitalization for HF, require specialist advisement.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Wait time 1 | At week three following study entry.
  The time between date referral made and date acknowledged by cardiologist.
Wait time 2 | At week sixteen following study entry.
  The time from acceptance for a procedure to time of pre-procedure imaging.
Wait time 3 | At week sixteen following study entry.
  The time from acceptance for a procedure to time of procedure.

SECONDARY OUTCOMES:
Morbidity 1 | At 30 days post procedure.
  Morbidity = all cause hospitalization and heart failure hospitalization post procedure.
Morbidity 2 | At one year post procedure.
  Morbidity = all cause hospitalization and heart failure hospitalization post procedure.
Mortality 1 | At 30 days post procedure.
  Mortality = all cause mortality
Mortality 2 | At one year post procedure.
  Mortality = all cause mortality

OTHER OUTCOMES:
Electronic referral patient experience survey | At day one (study entry).
  A survey of patient experience and satisfaction with the electronic referral method.
  Comments:
  The survey will be developed by the study investigator and each patient experience related question will be answered using the following scale: Strongly agree ☐ Agree ☐ Neither agree or disagree ☐ Disagree ☐ Strongly disagree. ☐ NA
Electronic referral usage - eReferrals answered | At day one (study entry).
  Proportion (%) of eReferral answered
Electronic referral usage - response time | At day one (study entry).
  median specialist response interval time (days).
Electronic referral usage - inappropriate eReferrals | At day one (study entry).
  proportion (%) of inappropriate eReferrals.
Electronic referral usage - specialist time | At day one (study entry).
  median time (hours) spent by specialist on eReferral.
Cost comparison 1 | At one day post procedure.
  Cost comparison between eReferral and traditional referrals based on number of baseline (pre-procedural) lab tests and investigations.
Cost comparison 2 | On the day prior to procedure.
  Cost comparison between eReferral and traditional referrals based on number of missed clinic visits.

CONTACTS AND LOCATIONS:
Locations (1):
- Kingston Health Sciences Centre, Kingston, Ontario, Canada